CLINICAL TRIAL: NCT06699940
Title: A Retrospective Registry Study to Evaluate Application of NeuroStar® Advanced Therapy for Depression and Comorbid Anxiety in Adolescents
Brief Title: A Retrospective Study to Evaluate NeuroStar® Advanced Therapy in Adolescents
Status: Completed | Type: Observational
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Other Study IDs: 20226718
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: MDD
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adolescent Cohort: Patients in TrakStar database between the age of 12-21 who received at least one TMS treatment.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Patients between the age of 12-21 received TMS treatment for MDD disorder.

SUMMARY:
To assess the real-world effectiveness of transcranial magnetic stimulation (TMS) for depression in large adolescent and young adult samples.

DETAILED DESCRIPTION:
This is a retrospective analysis. The purpose of this study is to collate real world data (RWD) from existing medical records of patients aged 12 to 21 years who received treatment with NeuroStar Advanced Therapy for Major Depressive Disorder (MDD) as determined by scores on the PHQ-9 and CGI-S assessment tool into a central registry database.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of Major Depressive Disorder (MDD), according to DSM-4/ICD-9 or DSM-5/ICD-10 criteria applicable on the date treatment with NeuroStar Advanced Therapy begins.
2. 12 to 21 years of age.
3. Male or female.
4. Treatment with NeuroStar Advanced Therapy.
5. Treatment start-date of November 1, 2008, or later.
6. Treatment end date on or before the date on which the retrospective study sample is extracted from the TrakStar database.
7. a) Per Protocol Subjects: Subject received a course of a minimum of 20 treatments with NeuroStar Advanced Therapy.

   b) Intent-to-Treat (ITT) Subjects: Subject received at least one treatment with NeuroStar Advanced Therapy.
8. Treatment with NeuroStar Advanced Therapy to the left dorsolateral prefrontal cortex (DLPFC) only.
9. Treatment with NeuroStar Advanced Therapy according to standardized NeuroStar Advanced Therapy treatment protocols of DASH and/or Standard per the current FDA clearance.
10. Each of GAD-7 and PHQ-9 scores available at each of pre-treatment (defined as the closest score available within 7 days prior to administration of the first treatment) and post-treatment (defined as the closest score available within ± 7 days of the date of the last treatment) evaluations for the single NeuroStar Advanced Therapy course.
11. Subjects with moderate or greater depression prior to NeuroStar Advanced Therapy (pre-treatment), defined as a score on the Physician Health Questionnaire-9 (PHQ-9) ≥ 10 within 7 days prior to the first treatment.

Exclusion Criteria:

- 1. Gap in NeuroStar Advanced Therapy treatment > 14 continuous days, where applicable.

2. More than one DLPFC treatment session on the same day.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between the age of 12-21 who were treated with NeuroStar Advanced Therapy for MDD on or after November 1, 2008 and the data was collected in TrakStar Database as standard of care practice
Sampling Method: Non-Probability Sample
Enrollment: 7690 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Efficacy Outcome | 8 weeks
  To assess the pre-treatment to post-treatment change in PHQ-9 scores for the adolescent patient population. PHQ-9 is the Patient Health Questionnaire is a 9-question patient-completed assessment. Total scores range from 0 to 27. Higher the score means higher the depression severity.

SECONDARY OUTCOMES:
Efficacy Outcome | 8 weeks
  To assess the pre-treatment to post-treatment change in CGI-S scores for the adolescent patient population. The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. The total score range from 1 to 7 where 1 is normal and 7 is extremely ill patient.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Cole, PhD, Study Director — Neuronetics
Locations (1):
- Neuronetics, Malvern, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Croarkin PE, Aaronson ST, Carpenter LL, Hutton TM, Pages K, Chen B, Sackeim HA. The Effectiveness of Transcranial Magnetic Stimulation in Adolescents and Young Adults With Major Depressive Disorder. JAACAP Open. 2025 Jul 1;3(4):1246-1258. doi: 10.1016/j.jaacop.2025.06.006. eCollection 2025 Dec. PMID 41367968